CLINICAL TRIAL: NCT01208194
Title: Phase 2, Randomized, Double-blind, Placebo-controlled, Multi-Center Study of a Maintenance Therapy With Immunomodulator MGN1703 in Patients With Advanced Colorectal Carcinoma With Disease Control After Initial First-line Therapy
Brief Title: Efficacy Study of a Maintenance Therapy With Immunomodulator MGN1703 in Patients With Advanced Colorectal Carcinoma
Acronym: IMPACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mologen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MGN1703-C02; 2009-017432-40 (EudraCT Number)
Record Dates: First submitted 2010-08-27; First posted 2010-09-23 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Advanced Colorectal Carcinoma
Keywords: Advanced colorectal carcinoma; Maintenance therapy; Immunomodulator
MeSH Terms: interventions — MGN1703; Immunologic Factors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MGN1703 (Experimental): Study medication
  Interventions: Drug: MGN1703
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MGN1703 — solution, 60 mg, twice a week, until progression
  Other Names: immunomodulator
  Arms: MGN1703
Drug: Placebo — solution, 60 mg, twice a week, until progression
  Arms: Placebo

SUMMARY:
This is a phase 2, randomized, double-blind, multi-center clinical study to evaluate efficacy and safety of a maintenance therapy with the immunomodulator MGN1703 compared to placebo control. The study will be conducted in patients with advanced colorectal carcinoma (AJCC Stage IV) with disease control after first-line standard chemotherapy regimens.

DETAILED DESCRIPTION:
The phase 2 study will be conducted in patients with advanced colorectal carcinoma with disease control after first-line standard chemotherapy regimens with oral or intravenous fluoropyrimidines/leucovorin and irinotecan or oxaliplatin combined with a standard dose of bevacizumab lasted between 4.5 and 6 months, whereas the treatment duration with irinotecan or oxaliplatin should not be less than 3 months. Studies confirmed that completely chemotherapy-free intervals can be applicable in patients with advanced colorectal carcinoma who achieved disease control after initial first-line chemotherapy. Those therapy holidays minimize toxicity and unnecessary treatment load, reduce intensity of treatment, allow patients to stay longer on therapy, prevent therapy discontinuations due to toxicity, preserve the ability to re-administer chemotherapy later, and increase quality of life of the patients. The therapy-free interval represents a possibility to evaluate the efficacy of the study drug, MGN1703.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects older than 18 years of age
* Histologically confirmed colorectal carcinoma
* Radiological confirmation of unresectable advanced colorectal carcinoma (AJCC Stage IV) prior to start of initial first-line therapy
* At least one measurable lesion according to RECIST measured within 2 weeks prior to treatment start in case of partial response or stable disease
* Prior initial first-line therapy included oral or intravenous fluoropyrimidines/leucovorin,irinotecan or oxaliplatin with or without a standard dose of bevacizumab lasted between 4.5 and 6 months and finished (last day of last cycle) within 2 weeks prior to treatment start (treatment duration with irinotecan or oxaliplatin should not be less than 3 months)
* Patients who achieved disease control measured as objective response or disease stabilization after initial first-line therapy
* No curative standard therapy is available for the patient after first-line treatment
* ECOG performance status 0-1
* Adequate organ function, hemoglobin ≥ 9 g/L, white blood cell count (WBC) ≥ 3.0 x 109/L, absolute neutrophil count ≥ 1.5 x 109/L, platelets > 100 x109/L, aspartate and alanine aminotransferase (AST and ALT) ≤ 2.5 x ULN, bilirubin < 1.5 x ULN, blood creatinine ≤ 1.5 X ULN, prothrombin time (PT) and activated thromboplastin time (aPTT) within normal range
* Negative pregnancy test in women with childbearing potential
* Expected adequacy of follow-up
* Signed informed consent form (ICF)

Exclusion Criteria:

* More than one line of systemic chemotherapy for metastatic colorectal carcinoma
* Tumor progression after initial first-line therapy
* Clinically significant concomitant diseases or conditions, which in opinion of the investigator would lead to an unacceptable risk for the subject to participate in the study
* Prior or current other malignancy, except adequately treated superficial bladder cancer, basal or squamous cell carcinoma of the skin or other cancer for which the subject has been disease free for more than 3 years
* Known central nervous system metastases
* Active or uncontrolled infections
* Transfusion-dependent anemia
* History of autoimmune disease or immune deficiency
* Known hypersensitivity to oligonucleotides or excipients of the formulation
* Pregnancy and/or nursing
* Concurrent chronic systemic immune therapy or immunosuppressant medication, including steroid treatment
* Concurrent chemotherapy, hormonal therapy (except hormonal contraception and hormonal replacement therapy for menopausal women), or immunotherapy within the last 2 weeks prior to randomization or during the conduct of the study - Concurrent radiotherapy within the last 6 months prior to randomization or during the conduct of the study
* Known HIV seropositivity or active hepatitis B or C infection
* Planned major surgery during the study
* Participation in another clinical study with other investigational drugs within 30 days prior to the first treatment day
* Vaccination within 3 months prior to the first treatment day
* Any medical, mental, psychological or psychiatric condition which in opinion of the investigator would not permit the subject to complete the study or understand the patient information
* Presence of drug and/or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of median progression-free survival (PFS) in both treatment groups | Measured on accrual time 3 years

SECONDARY OUTCOMES:
Assessment of PFS rate | Measured at landmarks 12, 18 and 24 weeks after treatment start, and afterwards every 6 weeks until treatment stop
Evaluation of median overall survival (OS) | Measured on accrual time 3 years
Assessment of OS proportion in both groups | Measured at landmarks 12, 18 and 24 weeks after treatment start, and afterwards every 6 weeks until treatment stop
Evaluation of overall response rate (ORR) | Measured on accrual time 3 years
Evaluation of duration of response (complete response, partial response, stable disease) as time from initial determination of response to progressive disease measured by RECIST | Measured on accrual time 3 years
Assessment of the dynamic of clinical and laboratory parameters | An average time: participants are followed until progress
Evaluation of immunologic response to MGN1703 | An average time: participants are followed until progress
Assessment of quality of life (QOL) | An average time: participants are followed until progress
Assessment of the safety profile of MGN1703 | An average time: participants are followed until progress

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Joachim Schmoll, Principal Investigator — Klinik für Innere Medizin IV, Universitätsklinikum Halle (Saale)
Locations (12):
- Klinik für Innere Medizin I, Abteilung für Klinische Onkologie, Medizinische Universität Wien, Vienna, Austria
- Oncology Clinic, Faculty Hospital Olomouc, Olomouc, Czechia
- Service de Cancérologie Digestive, Institut de Cancérologie Gustave Roussy, Villejuif, France
- Germany (6):
  - Onkologischer Schwerpunkt am Oskar-Helene-Heim, Berlin
  - Klinik für Innere Medizin IV, Onkologie/ Hämatologie/ Hämostaseologie, Universitätsklinikum Halle (Saale), Halle
  - Kath. Marienkrankenhaus GmbH, Allgemeine Onkologie, Hamburg
  - Schwerpunktpraxis für Hämatologie und Onkologie, Magdeburg
  - Klinik für Innere Medizin, Klinik für Hämatologie, Onkologie, Immunologie, Universitätsklinikum Giessen und Marburg GmbH, Marburg
  - Medizinische Klinik, Abteilung für Onkologie, Hämatologie Immunologie, Rheumatologie und Pulmologie Universität Tübingen, Immuntherapie, Station 65 Med. Klinik Abt. II, Tübingen
- Russia (2):
  - State Institution "Russian Scientific Oncology Center named after N.N. Blokhin RAMN", Moscow
  - Non-state health care institution "Central Clinical Hospital No. 2 named after N.A. Semashko OAO "RZHD", Moscow
- Mount Vernon Cancer Centre, Northwood, Middlesex, United Kingdom